CLINICAL TRIAL: NCT04138043
Title: A Phase 1, Randomised, Double-blind, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Subcutaneous Doses of GSK2330811 in Healthy Japanese Participants
Brief Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics of GSK2330811 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 208564
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Results first posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Healthy Volunteers
Keywords: GSK2330811; Healthy participants; Japanese; Pharmacokinetics; Safety; Subcutaneous dose

STUDY DESIGN:
Intervention Model Description: This is a parallel group study. Participants will be randomized to receive either GSK2330811 (450 mg) or placebo in an approximate ratio of 7:3.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSK2330811 450 mg (Experimental): Participants will receive a single 450 mg SC dose of GSK2330811, administered as three separate SC injections of 150 milligrams per milliliter [mg/mL]).
  Interventions: Drug: GSK2330811
- Placebo (Placebo Comparator): Participants will receive GSK2330811 matching placebo administered as three separate SC injections.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo is 0.9 percent sodium chloride solution. It will be administered as SC injection to abdomen by study personnel. Three injections will be used to match active doses.
  Arms: Placebo
Drug: GSK2330811 — GSK2330811 will be available as SC injection 150 mg/mL.
  Arms: GSK2330811 450 mg

SUMMARY:
This is a randomized, double-blind (sponsor-open), placebo-controlled, single-center study involving Japanese participants. The purpose of the study is to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity after a single subcutaneous (SC) dose of GSK2330811 in healthy Japanese participants. GSK2330811 is a humanized immunoglobulin G1 (IgG1) monoclonal antibody that binds and inhibits the action of Oncostatin M (OSM) and is being developed for the treatment of Crohn's disease (CD) and Systemic sclerosis (SSc). Participants will be randomized to receive either GSK2330811 (450 milligram [mg]) or placebo in an approximate ratio of 7:3.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests and 12-lead ECGs.
* A participant with a clinical abnormality or laboratory parameters outside the reference range for the healthy population being studied that is not specifically listed in the inclusion or exclusion criteria may be included if the investigator and sponsor medical monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or interpretation.
* Participants with body weight >=45 kilogram (kg) and body mass index (BMI) within the range 18.5-29.9 kg per square meter.
* Male participants.
* Participants capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Participants with Japanese ancestry, defined as having been born in Japan, being descendants of four ethnic Japanese grandparents and two ethnic Japanese parents, holding a Japanese passport or identity papers, and being able to speak Japanese. Participants should have lived outside Japan for less than 10 years at the time of screening.

Exclusion Criteria:

* Participants with sensitivity to any of the study treatments or components there of (including humanized monoclonal antibodies) or history of severe post treatment hypersensitivity reactions including erythema multiforme major, linear immunoglobulin A (IgA) dermatosis, toxic epidermal necrolysis and exfoliative dermatitis.
* Participants with any other history of significant allergy that in the opinion of the investigator contraindicates their participation in this study.
* Participants with an active infection or a history of serious infections as follows: Use of antimicrobials (antibacterials, antivirals, antifungals or antiparasitic agents) for an infection within 30 days prior to Day 1. Topical treatments may be allowed at the Investigator's discretion (in consultation with the Medical Monitor); A history of opportunistic or recurrent infections, as determined by the investigator; Currently active or unresolved infection (participants with 'trivial' infections such as tinea pedis may be eligible at the discretion of the investigator); Symptomatic herpes zoster within 3 months prior to screening; History of tuberculosis (TB) (active or latent) irrespective of treatment status; and a positive diagnostic TB test at screening (defined as a positive QuantiFERON test).
* Participants with any planned major surgical procedure during the study.
* Participants with a history of hematological disease, for example (but not limited to): significant anemia, platelet disorders including drug-induced thrombocytopenia or primary immune thrombocytopenia and coagulation disorders including von Willebrand's disease.
* Participants with a history of carcinoma in situ and malignant disease, with the exception of adequately treated non-metastatic basal or squamous cell cancer of the skin that has been fully treated and shows no evidence of recurrence after 3 years.
* Participants with QTc >450 millisecond (msec) at screening.
* Participants with use of prescription or non-prescription drugs (including recreational drugs and herbal medications) within 7 days or 5 half-lives (whichever is longer) prior to Day 1 unless in the opinion of the investigator (in consultation with the sponsor medical monitor) the medication will not interfere with the study or compromise participant safety. Paracetamol at doses of <=4 grams per day, and occasional use of non-steroidal anti-inflammatory drugs (NSAIDs) at licensed doses, are permitted.
* Participants who received live vaccination within 4 weeks prior to Day 1, or any plan to receive a live vaccination during the study (up to and including to the last follow-up visit).
* Participation in a clinical trial and has received an investigational medicine product (IMP) within the following time period prior to Day 1: 3 months, 5 half-lives, or twice the duration of the biological effect of the IMP (whichever is longer).
* Participants with exposure to more than 4 new chemical entities within 12 months prior to Day 1.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 3 months.
* Participants with platelet count or hemoglobin below the normal range at any time during screening.
* Participants with alanine aminotransaminase (ALT) >1.5 times upper limit of normal (ULN) at any time during screening.
* Participants with bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent) at any time during screening.
* Participants with presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb), or positive hepatitis C virus (HCV) antibody result at screening. Participants with positive HCV antibody due to prior resolved disease can be enrolled only if a confirmatory negative HCV Ribonucleic acid (RNA) test is obtained.
* Participants with positive human immunodeficiency virus (HIV) antibody test at screening.
* Participants with positive pre-study drug or alcohol screen.
* Participants with history of regular alcohol consumption within 6 months of the screening visit in excess of an average weekly intake of >21 units. One unit is equivalent to 8 gram of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Participants planning to travel to regions of high endemic infection, as determined by the investigator, for the duration of the study.
* Participants with unstable lifestyle factors, to the extent that in the opinion of the investigator they would interfere with the ability of a participant to complete the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male participants of 18 to 65 years of age at the time of signing the informed consent are inclusive.
Enrollment: 9 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, placebo-controlled, single-center study with single subcutaneous (SC) dose of GSK2330811 administered in healthy male Japanese participants.
Pre-assignment Details: A total of 9 participants were randomized and enrolled in this study.
Groups:
- Placebo: Participants received a single SC dose of Placebo, administered as three separate SC injections.
- GSK2330811 450 mg: Participants received a single 450 milligram (mg) SC dose of GSK2330811, administered as three separate SC injections of 150 milligrams per milliliter [mg/mL]).
Period: Overall Study
Arm/Group | Placebo | GSK2330811 450 mg
Started | 2 | 7
Completed | 2 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK2330811 450 mg | Total
Number analyzed (Participants) | 2 | 7 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.0 (2.83) | 29.1 (6.52) | 27.3 (6.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 7 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Japanese Heritage | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment. Safety Population consisted of all randomized participants who received at least one dose of study treatment.
Time Frame: Up to Day 126
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330811 450 mg
Number analyzed (Participants) | 2 | 7
Participants
  AEs | 2 | 6
  SAEs | 0 | 0

2. Primary Outcome: Number of Participants With Worst Case Vital Sign Results Relative to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Vital signs were measured in semi-supine position after 5 minutes of rest and included systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR). Participants were counted in the worst case category that their value changed to low, within range or high, unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the "Within Range or No Change" category. Participants were counted twice if values changed 'To Low' and 'To High', so the percentages were not added up to 100 percent (%). Participants with missing Baseline values were assumed as within range value. PCI ranges were: SBP (lower: <85, upper: >160 millimeter of mercury [mmHg]); DBP (lower: <45, upper: >100 mmHg); HR (lower: <40, upper: >110 beats per minute). Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment.
Time Frame: Baseline (Pre-dose, Day 1) and up to Day 126
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330811 450 mg
Number analyzed (Participants) | 2 | 7
Participants
  SBP, To low | 0 | 0
  SBP, To Within Range or No Change | 2 | 7
  SBP, To high | 0 | 0
  DBP, To low | 0 | 0
  DBP, To Within Range or No Change | 2 | 7
  DBP, To high | 0 | 0
  HR, To low | 0 | 0
  HR, To Within Range or No Change | 2 | 7
  HR, To high | 0 | 0

3. Primary Outcome: Change From Baseline in Body Temperature
Description: Body temperature was measured in semi-supine position after 5 minutes of rest for the participants in a quiet setting without distractions. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Pre-dose, Day 1), Day 1: 1, 4, 8 hours; Days 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 84 and 126
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Placebo | GSK2330811 450 mg
Number analyzed (Participants) | 2 | 7
Degrees Celsius
  Day 1: 1 hour, n=2,7 | 0.15 (0.212) | 0.06 (0.237)
  Day 1: 4 hour, n=2,7 | 0.40 (0.283) | 0.07 (0.287)
  Day 1: 8 hour, n=2,7 | 0.45 (0.071) | 0.40 (0.346)
  Day 2: n=2,7 | -0.15 (0.919) | -0.03 (0.486)
  Day 3: n=2,7 | -0.30 (0.283) | -0.34 (0.336)
  Day 5: n=2,7 | 0.20 (0.424) | -0.06 (0.800)
  Day 7: n=2,7 | -0.30 (0.566) | 0.09 (0.521)
  Day 10: n=2,7 | -0.10 (0.283) | -0.10 (0.862)
  Day 14: n=2,7 | 0.25 (0.495) | 0.21 (0.537)
  Day 21: n=2,7 | 0.05 (0.212) | 0.09 (0.609)
  Day 28: n=2,7 | 0.20 (0.424) | -0.06 (0.670)
  Day 42: n=2,7 | -0.60 (0.283) | -0.10 (0.695)
  Day 56: n=2,6: number analyzed (Participants) | 2 | 6
  Day 56: n=2,6 | 0.00 (0.141) | -0.03 (0.715)
  Day 84: n=1,6: number analyzed (Participants) | 1 | 6
  Day 84: n=1,6 | 0.90 (NA) — Standard deviation could not be calculated for single participant. | 0.30 (0.494)
  Day 126: n=0,6: number analyzed (Participants) | 0 | 6
  Day 126: n=0,6 |  | 0.28 (0.595)

4. Primary Outcome: Number of Participants With Worst Case Abnormal Electrocardiogram (ECG) Findings
Description: 12-lead ECGs were recorded in semi-supine position using an ECG machine. Number of participants with worst-case clinically significant and not clinically significant abnormal ECG findings have been presented. Clinically significant abnormal laboratory findings were those which were not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to Day 126
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330811 450 mg
Number analyzed (Participants) | 2 | 7
Participants
  Abnormal - not clinically significant | 0 | 1
  Abnormal - clinically significant | 0 | 0

5. Primary Outcome: Number of Participants With Maximum Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or Higher Clinical Chemistry Parameters
Description: Blood samples were collected for the analysis of clinical chemistry parameters. Clinical chemistry parameters were summarized according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0: Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening or disabling. Higher grade indicates more severity. Clinical chemistry parameters included: total bilirubin, calcium, creatinine and triglycerides.
Time Frame: Up to Day 126
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330811 450 mg
Number analyzed (Participants) | 2 | 7
Participants
  Total Bilirubin, Grade 1 | 0 | 1
  Total Bilirubin, Grade 2 | 0 | 0
  Total Bilirubin, Grade 3 | 0 | 0
  Total Bilirubin, Grade 4 | 0 | 0
  Calcium, Grade 1 | 2 | 5
  Calcium, Grade 2 | 0 | 0
  Calcium, Grade 3 | 0 | 0
  Calcium, Grade 4 | 0 | 0
  Creatinine, Grade 1 | 0 | 1
  Creatinine, Grade 2 | 0 | 0
  Creatinine, Grade 3 | 0 | 0
  Creatinine, Grade 4 | 0 | 0
  Triglycerides, Grade 1 | 0 | 1
  Triglycerides, Grade 2 | 0 | 0
  Triglycerides, Grade 3 | 0 | 0
  Triglycerides, Grade 4 | 0 | 0

6. Primary Outcome: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of the following hematology parameters: hemoglobin (Hb), lymphocytes (Lympho), platelet count (PC), neutrophil count (Neutro) and White Blood Cell count (WBC). The laboratory parameters were graded according to NCI-CTCAE version 5.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Higher grade indicates more severity. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. An increase was defined as an increase in CTCAE Grade relative to Baseline Grade.
Time Frame: Baseline (Pre-dose, Day 1) and up to Day 126
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330811 450 mg
Number analyzed (Participants) | 2 | 7
Participants
  Hb, Anemia, increase to Grade 1 | 0 | 0
  Hb, Anemia, increase to Grade 2 | 0 | 0
  Hb, Anemia, increase to Grade 3 | 0 | 0
  Hb, Anemia, increase to Grade 4 | 0 | 0
  Hb, Hb increased, increase to Grade 1 | 0 | 0
  Hb, Hb increased, increase to Grade 2 | 0 | 0
  Hb, Hb increased, increase to Grade 3 | 0 | 0
  Hb, Hb increased, increase to Grade 4 | 0 | 0
  Lympho,Lympho count decreased, increase to Grade 1 | 0 | 3
  Lympho,Lympho count decreased, increase to Grade 2 | 1 | 0
  Lympho,Lympho count decreased, increase to Grade 3 | 0 | 0
  Lympho,Lympho count decreased, increase to Grade 4 | 0 | 0
  Lympho,Lympho count increased, increase to Grade 1 | 0 | 0
  Lympho,Lympho count increased, increase to Grade 2 | 0 | 0
  Lympho,Lympho count increased, increase to Grade 3 | 0 | 0
  Lympho,Lympho count increased, increase to Grade 4 | 0 | 0
  PC, PC decreased,increase to Grade 1 | 0 | 3
  PC, PC decreased,increase to Grade 2 | 0 | 2
  PC, PC decreased,increase to Grade 3 | 0 | 1
  PC, PC decreased,increase to Grade 4 | 0 | 0
  Neutro,Neutro count decreased,increase to Grade 1 | 0 | 0
  Neutro,Neutro count decreased,increase to Grade 2 | 0 | 1
  Neutro,Neutro count decreased,increase to Grade 3 | 0 | 0
  Neutro,Neutro count decreased,increase to Grade 4 | 0 | 0
  WBC,Leukocytosis, increase to Grade 1 | 0 | 0
  WBC,Leukocytosis, increase to Grade 2 | 0 | 0
  WBC,Leukocytosis, increase to Grade 3 | 0 | 0
  WBC,Leukocytosis, increase to Grade 4 | 0 | 0
  WBC,WBC decreased, increase to Grade 1 | 0 | 0
  WBC,WBC decreased, increase to Grade 2 | 0 | 1
  WBC,WBC decreased, increase to Grade 3 | 0 | 0
  WBC,WBC decreased, increase to Grade 4 | 0 | 0

7. Primary Outcome: Number of Participants With Worst Case Any Increase in Urinalysis Results Post-Baseline Relative to Baseline
Description: Urine samples were collected for analysis of blood, glucose, ketones and protein by a dipstick method. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters of urine glucose, protein, blood and ketones can be read as negative (-), trace, 1+, 2+, 3+ indicating proportional concentrations in the urine sample. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Any increase means any increase to trace, 1+, 2+ or 3+ post-Baseline relative to Baseline. Number of participants with worst case any increase in urinalysis results post-Baseline relative to Baseline has been presented.
Time Frame: Baseline (Pre-dose, Day 1) and up to Day 126
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330811 450 mg
Number analyzed (Participants) | 2 | 7
Participants
  Blood | 1 | 1
  Glucose | 0 | 0
  Ketones | 0 | 1
  Protein | 1 | 2

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) for GSK2330811
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK2330811. PK parameters were calculated using standard non-compartmental analysis. Pharmacokinetic Population consisted of all participants in the Safety population who received at least one active dose of study treatment and had at least 1 non-missing PK assessment.
Time Frame: Day 1: Pre-dose, 8 hours; Days 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 84 and 126
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | GSK2330811 450 mg
Number analyzed (Participants) | 7
Nanogram per milliliter | 63259.308 (14.9290)

9. Secondary Outcome: Area Under the Plasma Concentration Time-curve From Time Zero to Infinity (AUC[0-infinity]) for GSK2330811
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK2330811. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: Day 1: Pre-dose, 8 hours; Days 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 84 and 126
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | GSK2330811 450 mg
Number analyzed (Participants) | 7
Hours*nanogram per milliliter | 45371065.201 (22.1925)

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC[0-t]) for GSK2330811
Description: as for outcome 9
Time Frame: Day 1: Pre-dose, 8 hours; Days 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 84 and 126
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | GSK2330811 450 mg
Number analyzed (Participants) | 7
Hours*nanogram per milliliter | 43157791.065 (22.8839)

11. Secondary Outcome: Apparent Systemic Clearance (CL/F) for GSK2330811
Description: as for outcome 9
Time Frame: Day 1: Pre-dose, 8 hours; Days 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 84 and 126
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | GSK2330811 450 mg
Number analyzed (Participants) | 7
Liter per hour | 0.010 (22.1925)

12. Secondary Outcome: Time to Cmax (Tmax) for GSK2330811
Description: as for outcome 9
Time Frame: Day 1: Pre-dose, 8 hours; Days 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 84 and 126
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2330811 450 mg
Number analyzed (Participants) | 7
Hours | 143.380 [94.82 to 216.25]

13. Secondary Outcome: Terminal Half-life (t1/2) for GSK2330811
Description: as for outcome 9
Time Frame: Day 1: Pre-dose, 8 hours; Days 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 84 and 126
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK2330811 450 mg
Number analyzed (Participants) | 7
Hours | 469.117 (14.8081)

14. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss/F) for GSK2330811
Description: as for outcome 9
Time Frame: Day 1: Pre-dose, 8 hours; Days 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 84 and 126
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | GSK2330811 450 mg
Number analyzed (Participants) | 7
Liter | 6.713 (12.2891)

15. Secondary Outcome: Number of Participants With Positive Anti-GSK2330811 Antibodies
Description: Serum samples were analyzed for the presence of anti-GSK2330811 antibodies using an antibody binding assay. The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for the specificity using the confirmation assay. Number of participants with confirmed positive anti-GSK2330811 antibodies are presented.
Time Frame: Up to Day 126
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330811 450 mg
Number analyzed (Participants) | 2 | 7
Participants | 0 | 0

16. Secondary Outcome: Platelet Count Nadir for GSK2330811
Description: Blood samples were collected at indicated time points for analysis of platelet count nadir for GSK2330811. Nadir was defined as the lowest post-Baseline value of the platelet count.
Time Frame: Days 1, 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 84 and 126
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Placebo | GSK2330811 450 mg
Number analyzed (Participants) | 2 | 7
Giga cells per liter | 211.5 (27.58) | 79.1 (29.48)

17. Secondary Outcome: Time to Platelet Count Nadir for GSK2330811
Description: Blood samples were collected at indicated time points for analysis of platelet count nadir for GSK2330811. Nadir was defined as the lowest post-Baseline value of the platelet count. Time to nadir was defined as Study Day of Nadir minus 1.
Time Frame: Days 1, 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 84 and 126
Population: Safety Population.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | GSK2330811 450 mg
Number analyzed (Participants) | 2 | 7
Days | 44.0 [4 to 84] | 20.0 [20 to 26]

18. Secondary Outcome: Hemoglobin Nadir for GSK2330811
Description: Blood samples were collected at the indicated time points for analysis of hemoglobin nadir for GSK2330811. Nadir was defined as the lowest post-Baseline value of the hemoglobin.
Time Frame: Days 1, 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 84 and 126
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK2330811 450 mg
Number analyzed (Participants) | 2 | 7
Grams per liter | 136.0 (8.49) | 134.9 (6.69)

19. Secondary Outcome: Time to Hemoglobin Nadir for GSK2330811
Description: Blood samples were collected at indicated time points for analysis of hemoglobin nadir for GSK2330811. Nadir was defined as the lowest post-Baseline value of the hemoglobin. Time to nadir was defined as Study Day of Nadir minus 1.
Time Frame: Days 1, 2, 3, 5, 7, 10, 14, 21, 28, 42, 56, 84 and 126
Population: Safety Population.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | GSK2330811 450 mg
Number analyzed (Participants) | 2 | 7
Days | 30.5 [20 to 41] | 55.0 [14 to 125]

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs and non SAEs were collected up to Day 126
Description: Safety Population consisted of all randomized participants who received at least one dose of study treatment.
Arm/Group | Placebo | GSK2330811 450 mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/7
Other Adverse Events (participants affected / at risk) | 2/2 | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2) | GSK2330811 450 mg (N=7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT04138043/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT04138043/SAP_001.pdf